CLINICAL TRIAL: NCT06586476
Title: A Randomized Clinical Trial to Investigate the Efficacy and Feasibility of Timed Awakening in the Treatment of Enuresis
Brief Title: The Role of Timed Awakening in Treatment of Enuresis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Evalynn Vasquez, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHLA-23-00080
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Nocturnal Enuresis; Voiding Dysfunction
Keywords: Lifting; Incontinence; Bedwetting
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Lifting

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard of care, which includes in-clinic urotherapy at evaluation and 30-minutes psychotherapy sessions (every 3 weeks).
- Nightly Timed Awakening (Experimental): Control-arm therapy plus a nightly timed-awakening intervention.
  Interventions: Behavioral: Nightly Timed Awakening

INTERVENTIONS:
Behavioral: Nightly Timed Awakening — Patients in this arm will be awakened 1-hr after going to bed by their caregiver(s) to use the restroom and then returned to sleep. This awakening will occur every night.
  Other Names: Lifting
  Arms: Nightly Timed Awakening

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of nightly timed awakening in the treatment of nocturnal enuresis in children aged 6-17. The main questions it aims to:

* Determine feasibility of nightly timed awakenings
* Determine the role, if any, of comorbidities on resolution of enuresis
* Determine incidence of daytime accidents
* Obtain patient and parental satisfaction scores

Researchers will compare a control group to treatment groups to see if there is any impact on nocturnal enuresis.

Participants will be woken up by parents in the middle of the night to use the restroom. In addition, participants will receive 30 minute psychotherapy sessions using telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Our inclusion criteria are new and recently evaluated (within past 6 months) patients who are English-speaking
* aged 6-17
* referred to the urology clinic for enuresis (Enuresis in our study is defined as nocturnal or diurnal enuresis (more than 1 bedwetting episode/week) for greater than 3 months)

Exclusion Criteria:

* Diagnosis of enuresis with comorbid diagnosis of diabetes mellitus (type 1 and 2), diabetes insipidus, chronic kidney disease, polyuria and/or polydipsia
* Structural urologic disease (evaluated via baseline imaging)
* Diagnosis of neurodevelopmental delays or conditions (i.e. celebral palsy, autism spectrum disorder) that hinders inability to follow age-appropriate instructions
* Not potty trained
* Improved or resolved enuresis for patients recently evaluated (within the past 6 months)
* Non-English speaking
* Patients currently on any over-active-bladder (OAB) medications (b3- agonists, antichloingerics) or alpha blockers for urinary symptoms (i.e. alfuzosin, tamsulosion, etc) or anti-diurectic medications for urinary symptoms (i.e.: desmopression (DDAVP))
* Patients currently using bed-wetting alarms
* Patients and families who are actively seeing Pediatric Clinical Urologic Psychologist.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent or participate in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of wet nights reported in electronic survey weekly for 12-weeks | Baseline to 12-weeks
  All study participants will report bed wetting via redcap electronic survey 1x/week for a 12-week period.

SECONDARY OUTCOMES:
Mean change from baseline in the number of wet nights/week reported in electronic survey | Baseline to 12-weeks
  All study participants will report bed wetting via redcap electronic survey 1x/week for a 12-week period.
Percentage of patients with increased number of wet nights at 24-week follow-up as reported in electronic survey. | 24-weeks post-intervention
  All study participants will report bed wetting via redcap electronic survey 24-week after completion of intervention
Mean number of nights reported weekly in electronic survey with timed awakening for 12-week period for intervention arm. | Baseline to 12-weeks
  Intervention arm will report bed wetting via redcap electronic survey 1x/week for a 12-week period.
Mean number of daytime accidents/week at baseline, end of 12-weeks and 24-weeks follow-up. | Baseline to 24-week follow-up
  All study participants will report bed wetting via redcap electronic survey 24-week after completion of intervention
Mean satisfaction score obtained from patient and parental satisfaction questionnaire. | Baseline to 12-weeks
  Mean Patient and Parental Satisfaction Scores (Pq-EnU behavioral sub-score) will be collected via telehealth sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Evalynn Vasquez, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No